CLINICAL TRIAL: NCT02782871
Title: A Randomised Control Trial to Compare the Pneupac VR1 Portable Ventilator and Manual Ven-tilation Via a Mapleson C- Circuit During the Intra-hospital Transfers of Intubated Patients
Brief Title: RCT: Compare - Pneupac VR1 to Manual Ventilation in Intubated Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Collaborators: St Thomas' Hospital, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GSTT 2016
Record Dates: First submitted 2016-05-22; First posted 2016-05-25 (Estimated); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: Transfer; Intra-hospital; Ventilator; Manual ventilation; Head and neck surgery
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Manual ventilation with Mapleson C-circuit
- Intervention (Experimental): Pneupac VR1 portable ventilator
  Interventions: Device: Pneupac VR1

INTERVENTIONS:
Device: Pneupac VR1 — A portable mechanical ventilator/resuscitator for medical personnel in the hospital, ambu-lance, fire, and police services.
  Arms: Intervention

SUMMARY:
Following major head and neck surgery it may be necessary to keep patients intubated and ventilated for at least 12 hours to allow the swelling associated with the operation to subside. Therefore patients (participants) are transferred to the intensive care unit anaesthetised, in-tubated and ventilated. Current practice is that patients are manually ventilated, by hand, during transfer from the operating theatre to the intensive care unit.

DETAILED DESCRIPTION:
Following major head and neck surgery it may be necessary to keep patients intubated and ventilated for at least 12 hours to allow the swelling associated with the operation to subside. Therefore patients (participants) are transferred to the intensive care unit anaesthetised, in-tubated and ventilated. Current practice is that patients are manually ventilated, by hand, during transfer from the operating theatre to the intensive care unit.

Studies show that use of manual ventilation causes variability in respiratory parameters and blood gas values due to inconsistent ventilation. A study in 2003 found that portable ventila-tor provided more consistent ventilation and patients were less likely to have a disparity in their blood gases, oxygenation and ventilation.. However, conventional ventilators are bulky, heavy, expensive and few and far between in the hospital and, in particular, the pre-hospital setting. The Pneupac VR1 ventilator is simple to use, small, portable and durable. It is easy to clean, low cost, light weight and magnetic resonance imaging (MRI) compatible.

The study will aim to directly compare the efficiency and efficacy (ventilation rate and tidal volumes) of manual ventilation against a new device, VR-1 portable ventilator, by Smith-Medical. The device is CE approved. The RCT will compare the efficacy and efficiency during transfer of the patient from theaters to intensive care in our establishment. The endpoint will be arrival to the intensive care unit (ICU) and transfer onto the ICU ventilator. This will be measured by collecting the pCO2, taken from an already in-situ arterial blood gas (ABG), at two time points - (a) just before patient transfer from theaters to the intensive care unit and (b) upon arrival at the intensive care unit and just prior to transfer onto the ITU ventilator.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Elective surgery
* ASA 1-3
* Undergoing Head and neck surgery, where routine care includes intubation, arterial line and post-operative transfer to intensive care unit intubated .
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:
* Have refused consent to participate in trial
* Emergency surgery
* Those patients who do not require intubation, arterial line and/ or transfer to intensive care intubated as routine practice for type of surgery/ procedure being undertaken

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Pre- and post transfer partial pressure carbon dioxide measurements, from blood samples, taken from in-situ arterial line | Average (mean) 10 minutes
  The difference in pCO2 between patients in the control and the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Boston, Study Chair — Guy's & St Thomas' Foundation NHS Trust R&D Department

IPD SHARING:
Plan to Share IPD: No